CLINICAL TRIAL: NCT00700843
Title: Long-Term Follow-up of Ohio State University Medical Center (OSUMC) Bariatric Patients
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Bradley Needleman, Associate Professor, Ohio State University
Other Study IDs: 2008H0008
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: bariatric surgery; long term follow up; gastric partitioning surgery; Roux-en-Y gastric bypass surgery; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obtain long-term follow-up results for bariatric patients who underwent medical management or surgery for treatment of morbid obesity by Ohio State University Medical Center (OSUMC).

DETAILED DESCRIPTION:
The purpose of this study is to obtain long-term follow-up results for bariatric patients who underwent medical management or surgery for treatment of morbid obesity by Ohio State University Medical Center (OSUMC) surgeons during the late 1970s, 1980s, and 1990s. Our hypothesis is that surgical intervention for treatment of morbid obesity leads to sustained weight loss and decreased obesity-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Treated by OSUMC physicians for obesity
* Informed Consent

Exclusion Criteria:

* Informed consent not given

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who participated in the bariatric program at OSUMC ten or more years ago, including bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Failure to lose and maintain loss of > or equal to 50% of excess body weight will be considered failure of the bariatric surgery. | 10 or more years after surgery

SECONDARY OUTCOMES:
The need for additional surgical or other intervention for treatment of morbid obesity following bariatric surgery will be considered failure of the surgery. | 10 or more years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Needleman, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States